CLINICAL TRIAL: NCT01768117
Title: A Single-arm, Open-label Study To Describe The Safety, Tolerability, And Immunogenicity Of Bivalent Rlp2086 Vaccine In Laboratory Workers >=18 To < =65 Years Of Age
Brief Title: Study To Describe The Safety, Tolerability, And Immunogenicity Of Bivalent Rlp2086 Vaccine In Laboratory Workers ≥18 To ≤65 Years Of Age
Acronym: B1971042
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1971042
Record Dates: First submitted 2013-01-08; First posted 2013-01-15 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-11

CONDITIONS: Meningitis, Meningococcal, Serogroup B
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — factor H-binding protein, Neisseria meningitidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rLP2086 (Experimental)
  Interventions: Biological: rLP2086

INTERVENTIONS:
Biological: rLP2086 — 0.5 ml intramuscular injection of 120 microgram bivalent rLP2085 administered at 0, 2 and 6 months

SUMMARY:
This study will assess the safety, tolerability and immunogenicity of bivalent rLP2086 vaccine in laboratory workers ≥18 to ≤65 years of age administered on a Month 0, 2, and 6 schedule. The study will recruit laboratory personnel (inclusive of Pfizer staff) who work directly with pathogenic Neisseria meningitidis in the context of the bivalent rLP2086 vaccine development program. The study will provide descriptive safety and immunogenicity data following vaccination of these individuals with bivalent rLP2086 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory personnel (inclusive of Pfizer staff) who work directly with pathogenic Neisseria meningitidis in the context of the bivalent rLP2086 vaccine development program.
2. Male or female subject aged ≥18 to ≤65 years at the time of enrollment.
3. Negative urine pregnancy test.

Exclusion Criteria:

1. Subjects receiving any allergen immunotherapy with a nonlicensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
2. A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B cell function or those receiving immunosuppressive therapy. Subjects with terminal complement deficiency are excluded from participation in this study.
3. Significant neurological disorder or history of seizure (excluding simple febrile seizure).
4. Current chronic use of systemic antibiotics.
5. Received any investigational drugs, vaccines, or devices within 28 days before administration of the first study vaccination.
6. Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
7. Prior receipt of any vaccine specifically targeting fHBP or LP2086 antigens.
8. History of microbiologically proven disease caused by Neisseria meningitidis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Frontage Clinical Services (Formally ABR), Hackensack, New Jersey, United States

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991

RESULTS

PARTICIPANT FLOW:
Groups:
- rLP2086: Enrolled to receive on a 0, 2-, 6- month schedule
Period: Overall Study
Arm/Group | rLP2086
Started | 13
Completed | 7
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | rLP2086
Number analyzed (Participants) | 13
Age, Customized [Number; unit: participants]
  18- 40 years | 5
  Greater than (>) 40 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ)
Time Frame: 1 month after vaccination 3
Measure: Number; unit: participants
Arm/Group | rLP2086
Number analyzed (Participants) | 6
participants
  PMB80 [A22] 1:16 (N=6) | 6 [54.1 to 100.0]
  PMB2001 [A56] 1:8 (N=5) | 5 [47.8 to 100.0]
  PMB2948 [B24] 1:8 (N=6) | 6 [54.1 to 100]
  PMB2707 [B44] 1:8 (N=6) | 3 [11.8 to 88.2]

2. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Time Frame: Vaccination 1 up to 1 month after Vaccination 3
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086
Number analyzed (Participants) | 13
percentage of participants | 46.2

3. Secondary Outcome: Number of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer Level >= LLOQ
Time Frame: 1 month after vaccination (Vac) 1, 2, Immediately prior to vaccination 3
Measure: Number; unit: participants
Arm/Group | rLP2086
Number analyzed (Participants) | 6
participants
  1 month after Vac 1: PMB80 [A22] 1:16 (N=6) | 3 [11.8 to 88.2]
  1 month after Vac 2: PMB80 [A22] 1:16 (N=5) | 3 [22.3 to 95.7]
  Immediately prior to Vac 3: PMB80 [A22] 1:16 (N=6) | 4 [54.1 to 100.0]
  1 month after Vac 1: PMB2001 [A56] 1:8 (N=6) | 4 [4.3 to 77.7]
  1 month after Vac 2: PMB2001 [A56] 1:8 (N=6) | 6
  Immediately prior to Vac 3: PMB2001 [A56] 1:8(N=6) | 4
  1 month after Vac 1: PMB2948 [B24] 1:8 (N=6) | 6
  1 month after Vac 2: PMB2948 [B24] 1:8 (N=6) | 6
  Immediately prior to Vac 3: PMB2948 [B24] 1:8(N=6) | 5
  1 month after Vac 1: PMB2707 [B44] 1:8 (N=6) | 2
  1 month after Vac 2: PMB2707 [B44] 1:8 (N=6) | 3
  Immediately prior to Vac 3: PMB2707 [B44] 1:8(N=6) | 2

4. Secondary Outcome: Number of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer Level >= LLOQ For All 4 Primary Test Strains Combined
Time Frame: 1 month after vaccination 3
Measure: Number; unit: participants
Arm/Group | rLP2086
Number analyzed (Participants) | 5
participants | 3 [14.7 to 94.7]

5. Secondary Outcome: Number of Participants With 4-fold Increase in Serum Bactericidal Assay Using Human Complement (hSBA) Titer Level
Time Frame: 1 month after vaccination 3
Measure: Number; unit: participants
Arm/Group | rLP2086
Number analyzed (Participants) | 6
participants
  PMB80 [A22] (N=6) | 5 [35.9 to 99.6]
  PMB2001 [A56] (N=5) | 5 [47.8 to 100.0]
  PMB2948 [B24] (N=6) | 4 [22.3 to 95.7]
  PMB2707 [B44] (N=6) | 3 [11.8 to 88.2]

ADVERSE EVENTS:
Time Frame: AE reported from Vaccination 1 to 1 month after last administration of investigational product (bivalent rLP2086). SAE reported from Vaccination 1 to 6 months after last administration of investigational product (bivalent rLP2086)
Description: Events collected on case report form were reported.
Arm/Group | rLP2086
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | rLP2086 (N=13)
Eye Pain (Eye disorders) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Presyncope (Nervous system disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1/7
Chills (General disorders) | 1 — An occurrence of chills reported as a systemic event, was also reported as an AE.

LIMITATIONS AND CAVEATS:
Results of immunogenicity endpoints were reported in ''number'' and not in ''proportion'' as per team's input.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.